CLINICAL TRIAL: NCT06943300
Title: Comparison of Aerobic Training and Circuit Training on Body Mass Index, Physical Fitness, and Quality of Life in Healthy Children
Brief Title: Comparison of Aerobic Training and Circuit Training in Healthy Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/25/aniqa asif
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy Population
Keywords: Obesity; Physical Activity; Aerobic Training; Circuit Training; Body Mass Index; Quality of Life
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Circuit-Based Exercise

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial will be conducted, recruiting healthy children within a specific age range 8-12. This study will be conducted in the Leader's Lyceum School. Two experimental groups will be made. Participants will be randomly assigned to either an aerobic training group or a circuit training group. Non-probability convenient sampling technique will be used. The study will include the children from age 8 to 12, both genders, healthy children. Both programs will be implemented for a set duration of 12 weeks, with specific parameters regarding intensity, duration, and exercise types. The project will assess changes in BMI, physical fitness components (e.g., cardiovascular endurance, muscular strength, flexibility), and quality of life through validated measures, including Pediatric Quality of Life Generic Score 4.0 (PedsQL), Physical Fitness Test, Presidential Fitness test and BMI.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A: Experiment Group A (aerobic Group); Children will receive Aerobic training.
  Interventions: Other: Aerboic Training; Other: Circuit Training
- Group B (Experimental): Group B: Experiment Group B (circuit group); Children will receive Circuit training.
  Interventions: Other: Aerboic Training; Other: Circuit Training

INTERVENTIONS:
Other: Aerboic Training — Group A will perform Aerobic training exercises will be conducted 2 times per 12 weeks in which the warm up phase for 10 minutes. 30 minutes of aerobic exercise like walking, jogging, cycling, calisthenics, rhythmic exercises, continuous slow running, sit ups and cool down phase for stretching Phase 1: stretching of upper limb, trunk, lower limb muscles for 10 minutes. Phase 2: Individualized walking, jogging, cycling, rhythmic exercises, continuous slow running, sit ups Phase 3: Cool down exercise for 10 minutes.
Other: Circuit Training — The training program will consist of 10 types of resistance and aerobic exercise and will be done 2 times per week for 12 weeks. Specifically, the resistance exercise program comprises of push-up, squat, crunches, lunge and superman exercise. An aerobic exercise program comprises of light jumping, running on the spot, foot stamping, stepping and jumping jack. Phase 1: In Warm up period, dynamic stretching for 10 minutes. Phase 2: Resistance and aerobic exercise (push-up, squat, crunches, lunge and superman exercise, light jumping, running on the spot, foot stamping, stepping and jumping jack) Phase 3: In cool down period, static stretching for 10 minutes.

SUMMARY:
Childhood obesity is a growing concern, with potential consequences for long-term health. The number of obese children has increased more than tenfold in the last forty years. Over the course of their lifetimes, more and more young people worldwide will be exposed to obesity, which will hasten the onset of type 2 diabetes, fatty liver, and cardiovascular problems. Promoting physical activity in children is crucial for maintaining a healthy weight and improving overall well-being. Less than 30% of kids and teenagers worldwide fulfill the recommended daily minimum of 60 minutes of moderate to intense physical activity. Since that most children and adolescents spend a significant amount of time traveling to and from school or attending school, schools may be the best places for interventions. This project will investigate the effectiveness of two common exercise approaches, aerobic training and circuit training, on body mass index (BMI), physical fitness, and quality of life in healthy children.

A randomized controlled trial will be conducted, recruiting healthy children within a specific age range 8-12. This study will be conducted in the Leader's Lyceum School.Two experimental groups will be made. Participants will be randomly assigned to either an aerobic training group or a circuit training group. Non-probability convenient sampling technique will be used. The study will include the children from age 8 to 12, both genders, healthy children. Both programs will be implemented for a set duration of 12 weeks, with specific parameters regarding intensity, duration, and exercise types. The project will assess changes in BMI, physical fitness components (e.g., cardiovascular endurance, muscular strength, flexibility), and quality of life through validated measures, including Pediatric Quality of Life Generic Score 4.0 (PedsQL), Physical Fitness Test, Presidential Fitness test and BMI.

ELIGIBILITY:
Inclusion Criteria:

* ⦁ School Age Children from age 7-12 years

  * Both Genders, Male and Female
  * Healthy and fit children
  * Interventions should be given inside the premises of school
  * Children with normal range BMI: 13.3-24.1
  * Children with presidential fitness score at or above the 85th percentile
  * Children with Quality of Life score: minimum 50

Exclusion Criteria:

* ⦁ Any Children havig any mental condition: Depession or Anxiety

  * Visual, vestibular, or balance disorders in the preceding six months
  * Children with any orthotic devices
  * Children undertaking any previous aerobic or circuit training
  * Refusal of any child or parent to participate

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
Pediatric Quality of Life Generic Score 4.0 (PedsQL) | Baseline, 4th week, 8th week, 12th week
  The PedsQL 4.0 Generic Core Scales is a standardized tool used to measure health-related quality of life in children aged 2 to 18 years, through self-report and parent proxy-report. It includes 23 items across four domains-physical, emotional, social, and school functioning. Items are rated on a 5-point scale and converted to scores from 0-100, with higher scores indicating better quality of life.The PedsQL 4.0 has demonstrated high reliability, with Cronbach's alpha values typically above 0.70 for subscales and >0.90 for the total score. It also shows strong validity, effectively distinguishing between healthy children and those with chronic conditions, and is sensitive to changes over time-making it a reliable and valid tool for assessing pediatric quality of life.
Physical Fitness Test | Baseline, 4th week, 8th week, 12th week
  A physical fitness test evaluates key components of fitness such as cardiovascular endurance, muscular strength, muscular endurance, flexibility, and body composition. It helps assess overall physical health and performance. When standardized and properly administered, these tests are generally considered valid (accurately measure fitness components) and reliable (produce consistent results over time).
Presidential Fitness Test | Baseline, 4th week, 8th week, 12th week
  The Presidential Fitness Test was a U.S. school-based program designed to assess children's physical fitness through activities like sit-ups, push-ups, a mile run, and flexibility tests. It aimed to promote health and fitness in youth. It has moderate to good reliability and validity for measuring specific fitness components like strength and endurance. It was generally consistent when properly administered, but less valid as a health-focused tool due to its emphasis on performance over personal progress.
Body Mass Index | Baseline, 4th week, 8th week, 12th week
  The BMI chart classifies individuals based on their body mass index (BMI) into categories like underweight, normal weight, overweight, and obesity. While valid for large population assessments, it doesn't directly measure body fat and may misclassify individuals, such as athletes or older adults. It's reliable for general screening, but additional measures are needed for a more accurate assessment of individual health.

CONTACTS AND LOCATIONS:
Overall Officials: Aniqa Asif, MS-PPT, Principal Investigator — Riphah International University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmadi A, Moheb-Mohammadi F, Navabi ZS, Dehghani M, Heydari H, Sajjadi F, Khodarahmi S. The effects of aerobic training, resistance training, combined training, and healthy eating recommendations on lipid profile and body mass index in overweight and obese children and adolescents: A randomized clinical trial. ARYA Atheroscler. 2020 Sep;16(5):226-234. doi: 10.22122/arya.v16i5.1990. PMID 33889189